CLINICAL TRIAL: NCT05330325
Title: A Study Comparing the Effect and Safety of Once Weekly Dosing of Somapacitan With Daily Norditropin® as Well as Evaluating Long-term Safety of Somapacitan in a Basket Study Design in Children With Short Stature Either Born Small for Gestational Age or With Turner Syndrome, Noonan Syndrome, or Idiopathic Short Stature
Brief Title: A Research Study to Compare Somapacitan Once a Week With Norditropin® Once a Day in Children Who Need Help to Grow
Acronym: REAL 8
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN8640-4467; 2021-005607-13 (EudraCT Number); U1111-1270-0862 (Other: World Health Organization (WHO))
Record Dates: First submitted 2022-04-08; First posted 2022-04-15 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: SGA, Turner Syndrome, Noonan Syndrome, ISS
MeSH Terms: conditions — Turner Syndrome; Noonan Syndrome | interventions — somapacitan; Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Somapacitan (Experimental): Participants will receive Somapacitan for 273 weeks
  Interventions: Drug: Somapacitan
- Norditropin® (Active Comparator): Participants will receive Norditropin® for 52 weeks (main treatment period) and Somapacitan for 221 weeks (extension period)
  Interventions: Drug: Norditropin®

INTERVENTIONS:
Drug: Somapacitan — Somapacitan will be administered subcutaneously (s.c.) once weekly using PDS290 pen-injector.
  Arms: Somapacitan
Drug: Norditropin® — Norditropin® will be administered s.c. once daily using FlexPro® pen-injector.
  Arms: Norditropin®

SUMMARY:
The study compares two medicines for treatment of children born small and who stay small, or with Turner Syndrome, Noonan Syndrome, or idiopathic short stature. The purpose of the study is to see how well treatment with somapacitan works compared to treatment with Norditropin®. Somapacitan is a new medicine, and Norditropin® is a medicine doctors can already prescribe in some countries. The study will last for upto 5.5 years. The participants will either get somapacitan once a week up to 5.5 years or Norditropin® once a day for 1 year followed by somapacitan once a week for up to 4.5 years. Which treatment the participants get is decided by chance.

ELIGIBILITY:
Inclusion criteria:

1. Informed consent of parent or legally acceptable representative of participant and child assent, as age appropriate must be obtained before any study-related activities. Study-related activities are any procedures that are carried out as part of the study, including activities to determine suitability for the study.
2. No prior exposure to growth promoting therapy, including but not limited to growth hormone, IGF-I and ghrelin analogues.

   Applicable to children with SGA:
3. Born small for gestational age (birth length below -2 SDS OR birth weight below -2 SDS OR both) (according to national standards).
4. Prepubertal children:

   1. Boys:

      * Age above or equal to 2 years and 26 weeks and below 11.0 years at screening.
      * Testis volume below 4 mL
   2. Girls:

      * Age above or equal to 2 years and 26 weeks and below 10.0 years at screening.
      * Tanner stage 1 for breast development: No palpable glandular breast tissue)
5. Impaired height defined as at least 2.5 standard deviations below the mean height for chronological age and sex at screening according to the standards of Centers for Disease Control and Prevention.
6. Impaired height velocity defined as annualized height velocity below the 50th percentile for chronological age and sex according to the standards of Prader calculated over a time span of minimum 6 months and maximum 18 months prior to screening.
7. Body Mass Index below the 95th percentile according to Centers for Disease Control and Prevention, Body Mass Index-for-age growth charts.

   Applicable to girls with TS:
8. Confirmed diagnosis of TS by 30-cell (or more) lymphocyte chromosomal analysis.*
9. Prepubertal girls:

   * Age above or equal to 2 years and 26 weeks and below 10.0 years at screening.
   * Tanner stage 1 for breast development: No palpable glandular breast tissue)
10. Impaired height defined as at least 2.0 standard deviations below the mean height for chronological age and sex at screening according to the standards of Centers for Disease Control and Prevention.
11. Historical height measured 6-18 months prior to screening.
12. Thyroid hormone replacement therapy should be adequate and stable for at least 90 days prior to randomization, if applicable.

    Applicable to children with NS:
13. Clinical diagnosis of NS according to van der Burgt score list
14. Prepubertal children:

    1. Boys:

       * Age above or equal to 2 years and 26 weeks and below 11.0 years at screening.
       * Testis volume below 4 mL
    2. Girls:

       * Age above or equal to 2 years and 26 weeks and below 10.0 years at screening.
       * Tanner stage 1 for breast development: No palpable glandular breast tissue)
15. Impaired height defined as at least 2.0 standard deviations below the mean height for chronological age and sex at screening according to the standards of Centers for Disease Control and Prevention.
16. Historical height measured 6-18 months prior to screening.
17. Thyroid hormone replacement therapy should be adequate and stable for at least 90 days prior to randomization, if applicable.

    Applicable to children with ISS:
18. Prepubertal children:

    1. Boys:

       * Age above or equal to 2 years and 26 weeks and below 11.0 years at screening.
       * Testis volume below 4 mL
    2. Girls:

       * Age above or equal to 2 years and 26 weeks and below 10.0 years at screening.
       * Tanner stage 1 for breast development: No palpable glandular breast tissue)
19. Bone age:

    1. Boys:

       * Bone age below or equal to 12 years.
       * Bone age not delayed or advanced more than 2 years compared to chronological age.
    2. Girls:

       * Bone age below or equal to 11 years.
       * Bone age not delayed or advanced more than 2 years compared to chronological age.
20. Impaired height defined as at least 2.5 standard deviations below the mean height for chronological age and sex at screening according to the standards of Centers for Disease Control and Prevention.
21. Historical height measured 6-18 months prior to screening.
22. One normal GH secretion (GH peak above 7 ng/mL) during GH stimulation test performed within 18 months prior to screening or if such a test is not available for children with ISS, a test should be performed as part of the screening assessments and the result must be available prior to randomization.

    * If a 30-cell count is not available for patients with TS, a test should be done, and results must be available prior to randomization.

Exclusion criteria:

1. Known or suspected hypersensitivity to study intervention(s) or related products.
2. Previous randomization into same sub-study in this study.
3. Receipt of any investigational medicinal product within 3 months before screening or participation in another clinical study at the time of randomization.
4. Children with suspected or confirmed growth hormone deficiency according to local practice.
5. laboratory of

   1. fasting plasma glucose above or equal to 126 mg/dL (7.0 mmol/L) or
   2. HbA1c above or equal to 6.5%.
6. Current inflammatory diseases requiring systemic corticosteroid treatment for longer than 2 consecutive weeks within the last 3 months prior to screening.
7. Children requiring inhaled glucocorticoid therapy at a dose greater than 400 µg/day of inhaled budesonide or equivalent (i.e., 250 µg/day for fluticasone propionate) for longer than 4 consecutive weeks within the last 12 months prior to screening.
8. Concomitant administration of other treatments that may have an effect on growth, e.g., but not limited to methylphenidate for treatment of attention deficit hyperactivity disorder (ADHD).
9. Diagnosis of attention deficit hyperactivity disorder (ADHD).
10. History or known presence of any malignancy, intracranial tumour, or intracranial cyst.
11. History or known presence of active Hepatitis B or Hepatitis C (exceptions to this exclusion criterion is the presence of antibodies due to vaccination against Hepatitis B).
12. Any disorder, which in the investigator's opinion, might jeopardize participant's safety or compliance with the protocol.
13. The participant or the parent/legally acceptable representative is likely to be non-compliant in respect to study conduct, as judged by the investigator.
14. Current treatment with sex hormones or aromatase inhibitors.
15. Any known or suspected clinically significant abnormality likely to affect growth or the ability to evaluate growth with standing height measurements, such as, but not limited to:

    1. Known family history of skeletal dysplasia.
    2. Significant spinal abnormalities including but not limited to scoliosis, kyphosis and spina bifida variants.
    3. Any other disorder/condition that can cause short stature such as, but not limited to, psychosocial deprivation, nutritional disorders, chronic systemic illness and chronic renal disease.

Applicable to children with SGA:

1. TS (including mosaicism).
2. NS.
3. Hormonal deficiencies.
4. Children who are small due to malnutrition defined as -2 standard deviations according to standards. 0¬-5 years: weight for height on World Health Organization Multicentre Growth Reference Study 2006. Above 5 years: World Health Organization 2007 Body Mass Index.
5. Known chromosomal aneuploidy or significant gene mutations causing medical 'syndromes' with short stature, including but not limited to Laron syndrome, Prader-Willi syndrome, Russell-Silver Syndrome, skeletal dysplasias, abnormal SHOX gene analysis or absence of GH receptors.

Applicable to children with TS:

1. NS.
2. Mosaicism below 10%.
3. TS with Y-chromosome mosaicism where gonadectomy has not been performed.
4. NYHA class II or above or requiring medication for any heart condition.
5. Coeliac disease where participant is not stable on gluten free diet for the previous 12 months prior to screening.

Applicable to children with NS:

1. TS (including mosaicism).
2. Noonan-related disorders: Noonan syndrome with multiple lentigines (formerly called 'LEOPARD' syndrome), Noonan syndrome with loose anagen hair, cardiofaciocutaneous syndrome (CFC), Costello syndrome, neurofibromatosis type 1 (NF1) and Legius syndrome. Molecular genetic panel testing results must be available prior to randomisation to exclude these.
3. Coeliac disease where participant is not stable on gluten free diet for the previous 12 months prior to screening.

Applicable to children with ISS:

1. TS (including mosaicism).
2. NS.
3. Hormonal deficiencies.
4. Born small for gestational age (defined as birth length below -2 SDS OR birth weight below -2 SDS OR both) (according to national standards).
5. Known chromosomal aneuploidy or significant gene mutations causing medical 'syndromes' with short stature, including but not limited to Laron syndrome, Prader-Willi syndrome, Russell-Silver Syndrome, skeletal dysplasias, abnormal SHOX gene analysis or absence of GH receptors.

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 399 (Estimated)
Dates: Start 2022-08-10 (Actual); Primary Completion 2024-08-05 (Actual); Study Completion 2027-10-29 (Estimated)

PRIMARY OUTCOMES:
Height velocity reported separately for small for gestational age (SGA), Turner syndrome (TS), Noonan syndrome (NS) and idiopathic short stature (ISS) | From baseline (week 0) to visit 7 (week 52)
  Measured in centimeter per year (cm/year)

SECONDARY OUTCOMES:
Change in Height standard deviation scores (SDS) reported separately for SGA, TS, NS and ISS | From baseline (week 0) to visit 7 (week 52)
  Measured in score. Positive score indicates that the value is closer to or above the reference population compared to baseline.
Change in Height Velocity SDS reported separately for SGA, TS, NS and ISS | From baseline (week 0) to visit 7 (week 52)
  Measured in score. Positive score indicates that the value is closer to or above the reference population compared to baseline.
Change in bone age reported separately for SGA, TS and NS | From baseline (week 0) to visit 7 (week 52)
  Measured in ratio
Change in bone age for ISS | From screening (visit 1) to visit 7 (week 52)
  Measured in ratio
Change in insulin-like growth factor 1 (IGF-1) SDS reported separately for SGA, TS, NA and ISS | From baseline (week 0) to visit 7 (week 52).
  Measured in score. Positive score indicates that the value is closer to or above the reference population compared to baseline.
Change in insulin-like growth factor binding protein-3 (IGFBP-3) SDS reported separately for SGA, TS, NA and ISS | From baseline (week 0) to visit 7 (week 52).
  Measured in score. Positive score indicates that the value is closer to or above the reference population compared to baseline.
Change in fasting plasma glucose reported separately for SGA, TS, NS and ISS | From screening (visit 1) to visit 7 (week 52)
  Measured in millimoles per litre (mmol/L)
Change in homeostatic model assessment-B (HOMA-B) reported separately for SGA, TS, NS and ISS | From screening (visit 1) to visit 7 (week 52)
  Measured in percentage (%)
Change in homeostatic model assessment of insulin resistance (HOMAIR) reported separately for SGA, TS, NS and ISS | From screening (visit 1) to visit 7 (week 52)
  Measured in %
Change in glycated haemoglobin (HbA1c) reported separately for SGA, TS, NS and ISS | From screening (visit 1) to visit 7 (week 52)
  Measured in percentage of HbA1c
Weekly average somapacitan concentration (Cavg) based on population PK analysis | From visit 3 (week 4) to visit 7 (week 52)
  Measured in nanograms per milliliter (ng/mL)
Change in fasting plasma glucose reported separately for SGA, TS, NS and ISS | From screening (visit 1) to visit 15 (week 156)
  Measured in mmol/L
Change in homeostatic model assessment-B (HOMA-B) reported separately for SGA, TS, NS and ISS | From screening (visit 1) to visit 15 (week 156)
  Measured in %
Change in homeostatic model assessment of insulin resistance (HOMA-IR) reported separately for SGA, TS, NS and ISS | From screening (visit 1) to visit 15 (week 156)
  Measured in %
Change in glycated haemoglobin (HbA1c) reported separately for SGA, TS, NS and ISS | From screening (visit 1) to visit 15 (week 156)
  Measured in percentage of HbA1c

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency dept. 2834, Study Director — Novo Nordisk A/S
Locations (197):
- United States (35):
  - Univ of AL at Birmingham_BRM, Birmingham, Alabama
  - Children's Hospital Los Angeles - Endocrinology, Los Angeles, California
  - Sutter Valley Med Fdt Ped Endo, Sacramento, California
  - Rady Childrens Hosp San Diego, San Diego, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mt Ped and Endo, Centennial, Colorado
  - Ped Endo Assoc PC-G.V, Greenwood Village, Colorado
  - Nemours/AI duPont Hosp-Chld, Wilmington, Delaware
  - Childrens National Medical Ctr, Washington D.C., District of Columbia
  - Nemours Chld Clnc Jacksonville, Jacksonville, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - St. Luke's Children's Endo, Boise, Idaho
  - Rocky Mt Clin Res, LLC, Idaho Falls, Idaho
  - Riley Hosp for Child-Indiana U, Indianapolis, Indiana
  - University OF Iowa, Iowa City, Iowa
  - UMass Medical School, Worcester, Massachusetts
  - Univ of Minnesota M.C.H., Minneapolis, Minnesota
  - Children's Minnesota, Saint Paul, Minnesota
  - Univ of Mississippi Med Ctr, Jackson, Mississippi
  - The Children's Mercy Hospital, Kansas City, Missouri
  - Goryeb Children's Hospital, Morristown, New Jersey
  - UBMD Peds-Div of Endo/Diabetes, Buffalo, New York
  - NYU Langone Hospital-LI, Garden City, New York
  - NYU Langone Hospital-LI, Mineola, New York
  - WakeMed Childn Endo-Dbt_Raleig, Raleigh, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - CCHMC_Cinc, Cincinnati, Ohio
  - Univ Oklahoma Sci Ctr OK City, Oklahoma City, Oklahoma
  - UPMC Child Hosp-Pittsburgh, Pittsburgh, Pennsylvania
  - UT Southwestern Med Cntr, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
  - University Of Virginia Hospitl, Charlottesville, Virginia
  - MultiCare Inst for Res & Innov, Tacoma, Washington
  - Marshfield Clinic, Marshfield, Wisconsin
- Austria (4):
  - Kepler Universitätsklinikum GmbH - Med Campus IV (vorm.LFKK), Linz, Upper Austria
  - Krankenhaus der Stadt Dornbirn, Dornbirn
  - LKH St. Poelten, Kinder-und Jugendheilkunde, Sankt Pölten
  - Salzkammergut-Klinikum Vöcklabruck, Vöcklabruck
- Belgium (4):
  - UZ Brussel, Brussels
  - Cliniques Universitaires Saint-Luc - Serv. Pédiatrie, Brussels
  - UZA - UZ Antwerpen - Kinderziekenhuis, Edegem
  - UZ Leuven - Kindergeneeskunde, Leuven
- Brazil (4):
  - Centro de Diabetes Curitiba, Curitiba, Paraná
  - Santa Casa Sao Paulo, São Paulo, São Paulo
  - CPQuali Pesquisa Clínica Ltda, São Paulo, São Paulo
  - Centro de Pesquisa Clínica do Hospital das Clínicas da Faculdade de Medicina da USP, São Paulo, São Paulo
- Bulgaria (4):
  - UMHAT "Dr. Georgi Stranski" Pleven, Pleven
  - UMHAT Sveti Georgi EAD, Plovdiv, Clinic of Pediatrics, Plovdiv
  - SHATPD - Prof. Ivan Mitev EAD, Sofia
  - UMHAT Sveta Marina EAD, First Pediatric Clinic, Varna
- Children's Hosp-East Ontario, Ottawa, Ontario, Canada
- China (14):
  - Beijing Children's Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Liuzhou Maternity and Child Healthcare Hospital-Child Healthcare, Liuchow, Guangxi
  - Sanya Central Hospital (Hainan Third People's Hospital)-Pediatric, Sanya, Hainan
  - Henan Children's Hospital Zhengzhou Children's Hospital-Endocrine Genetics and Metabolism, Zhengzhou, Henan
  - Wuhan Children Hospital-Endocrine Genetics and Metabolism, Wuhan, Hubei
  - Wuhan Children Hospital, Wuhan, Hubei
  - Tongji Hospital, Tongji Medical College of HUST-Pediatric, Wuhan, Hubei
  - Hunan Children's Hospital-Child Health Center, Changsha, Hunan
  - The First Bethune Hospital of Jilin University-Pediatric, Changchun, Jilin
  - Shandong Provincial Hospital-Pediatric, Jinan, Shandong
  - Shanghai Children's Hospital -Endocrine Genetics and Metabolism, Shanghai, Shanghai Municipality
  - Shanghai Children's Medical Center-Endocrine Genetics and Metabolism, Shanghai, Shanghai Municipality
  - Chengdu Women's and Children's Central Hospital, Chengdu, Sichuan
- Croatia (2):
  - KBC "Sestre Milosrdnice", Zagreb
  - KBC Zagreb, Zavod za dječju endokrinologiju i dijabetes, Zagreb
- HUS Uusi lastensairaala, Helsinki, Finland
- France (12):
  - Centre Hospitalier Régional Universitaire d' Angers, Angers
  - Centre Hospitalier Universitaire D'Angers-2, Angers
  - Centre Hospitalier Universitaire de Bordeaux-Hopital Pellegrin, Bordeaux
  - CHU Pellegrin, Bordeaux
  - Ap-Hp-Hopital de Bicetre-1, Le Kremlin-Bicêtre
  - Hopital de Bicetre_Le Kremlin-Bicetre, Le Kremlin-Bicêtre
  - Assistance Publique Hopitaux de Marseille-Hopital de La Timone-2, Marseille
  - Hopital de La Timone, Marseille Cédex 05
  - Ap-Hp-Hopital Necker, Paris
  - Hôpital Necker, Paris
  - CHU de Toulouse, Toulouse
  - Hopital Des Enfants, Toulouse
- Germany (5):
  - Universitätsklinikum Bonn - Kinderklinik, Bonn
  - Universitätsklinikum Erlangen - Kinder- und Jugendklinik, Erlangen
  - Endokrinologikum Frankfurt, Frankfurt am Main
  - Klinik für Allgemeine Pädiatrie und Neonatologie, Homburg
  - Universität des Saarlandes - Pädiatrie und Neonatologie, Homburg
- Greece (7):
  - U.G.H. "Attikon", Pediatric Endocrinology Outpatient Clinic, Athens
  - Childrens' Hospital of Athens "Agia Sofia", Goudi/Athens
  - P & A Kyriakou Childrens' Hospital - Department of Endocrinology Growth and Development, Goudi/Athens
  - General University of Patra - Paediatric Department, Pátrai
  - 'Ippokrateio' General Hospital of Thessaloniki, Thessaloniki
  - "AHEPA" University General Hospital of Thessaloniki, Thessaloniki
  - Ippokrateio Gen Hosp of Thessaloniki, 1st Pediatric Clinic, Thessaloniki
- India (3):
  - Amrita Institute Of Medical Sciences & Research Centre, Kochi, Kerala
  - Jehangir Clinical Development Centre, Pune, Maharashtra
  - All India Institute of Medical Sciences, New Dehli, New Delhi
- Ireland (4):
  - Cork University Hospital, Cork
  - CHI at Temple Street, Dublin
  - CHI Crumlin Dept of Endocrinology, Dublin
  - CHI Tallaght University Hospital, Dublin
- Israel (5):
  - Soroka MC - Pediatric Endocrinology, Beersheba
  - Rambam MC - Department of Pediatrics A, Haifa
  - Schneider MC - Endrocrinology and Diabetes, Petah Tikva
  - Sheba MC - Pediatric endocrinology and adolescent diabetes clinics, Tel Litwinsky
  - Shamir MC - Pediatric and Adolescents Endocrinology unit, Ẕerifin
- Italy (9):
  - Ospedale San Raffaele S.r.l. - Unità Clinica Pediatria e neonatologia, Milan, Lombardy
  - IRCCS Meyer Firenze, Florence
  - Ospedale Pediatrico Gaslini, Genova
  - Ospedale San Raffaele UO di Pediatria e UO di Neonatologia, Milan
  - Università degli Studi della Campania "L. Vanvitelli", Napoli
  - Bambin Gesù, Roma
  - Ospedale Pediatrico Bambino Gesu, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome
  - Fondazione Policlinico Universitario Agostino Gemelli IRCS, Rome
- Japan (20):
  - Fukuoka Children's Hospital_Endocrinology and Metabolism, Fukuoka-shi, Fukuoka
  - Fukuoka Children's Hospital, Fukuoka-shi, Fukuoka
  - Hyogo Prefectual Kobe Children's Hospital Dept. Metab & endo, Kobe-shi, Hyogo
  - Hyogo Prefectual Kobe Children's Hospital_Metab & endo, Kobe-shi, Hyogo
  - Univ.HP, Kyoto Pref Univ of Medicine, Dept. of Pediatrics, Kyoto
  - Nara Prefecture General Medical Center_Nephrology, Nara-shi, Nara
  - Nara Prefecture General Medical Center, Nara-shi, Nara
  - Niigata University Medical & Dental Hospital_Pediatrics, Niigata-shi, Niigata
  - Okayama Medical Center_Cardiology, Okayama-shi, Okayama
  - Osaka City General Hospital, Pediatric Endocrinology and Me, Osaka
  - Osaka Women's and Children's Hospital, Osaka
  - Saitama Children's Medical Center, Endocrinorogy&Metabolism, Saitama-shi, Saitama
  - Hokkaido University Hospital, Pediatrics, Sapporo, Hokkaido
  - Hokkaido University Hospital_Pediatrics, Sapporo, Hokkaido
  - Shizuoka Children's Hospital, Department of Diabetes and metabolism, Shizuoka-shi, Shizuoka
  - Institute of Science Tokyo Hospital_Pediatrics, Tokyo
  - Institute of Science Tokyo Hospital, Tokyo
  - National Center for Child Health and Development_Endo and Metabo, Tokyo
  - Keio University Hospital_Pediatrics, Tokyo
  - Fujita Health University Hospital, Pediatrics, Toyoake, Aichi
- Children's Clinical University Hospital, Riga, Latvia
- Hospital of Lithuanian University of Health Sciences Kauno klinikos, Kaunas, Lithuania
- Malaysia (5):
  - Hospital Universiti Sains Malaysia_Kota Bharu, Kelantan, Kota Bharu, Kelantan
  - University Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur
  - University Malaya Medical Centre, Lembah Pantai, Kuala Lumpur
  - Hospital Al-Sultan Abdullah UiTM, Bandar Puncak Alam, Selangor
  - University Technology MARA (UiTM) - Puncak Alam, Bandar Puncak Alam Selangor Darul Ehsan
- Consultorio de Endocrinología y Pediatría, Puebla City, Mexico
- Erasmus MC, Rotterdam, Netherlands
- Poland (9):
  - Kliniczny Szpital Wojewodzki nr 2 im. Sw. Jadwigi Krolowej w Rzeszowie, Rzeszów, Podkarpackie Voivodeship
  - UCK, Klinika Pediatrii, Diabetologii i Endokrynologii,, Gdansk
  - Górnośląskie Centrum Zdrowia Dziecka Szpital Kliniczny Nr 6, Katowice
  - Uniwer. Szpital Dzieciecy Klinika Endokry. Dzieci i Mlodzie, Krakow
  - Uniwersytecki Szptal Dziecięcy w Krakowie, Krakow
  - Klinika Endokrynologii i Chorób Metabolicznych, Lodz
  - SPSK nr 1 im Prof. T Sokolowskiego, Szczecin
  - Klinika Pediatrii SUM, SPSK nr 1 im. prof.S.Szyszko w Zabrzu_LOC#1, Zabrze
  - SPSK nr 1 im. prof.S.Szyszko w Zabrzu, Zabrze
- Portugal (5):
  - Unidade Local de Saúde São José EPE- Hospital D. Estefânia, Lisbon
  - Centro Hospitalar Lisboa Norte, Lisbon
  - Unidade Local De Saude De Santa Maria E.P.E., Lisbon
  - Unidade Local de Saúde de Santo António, E.P.E, Porto
  - Centro Hospitalar de Vila Nova de Gaia, Vila Nova de Gaia
- Saudi Arabia (2):
  - King Faisal Specialist Hospital & Research Centre, Riyadh, Riyadh
  - National Guard Hospital, Riyadh
- Serbia (6):
  - University Clinical Centre Nis, Niš, RS
  - University Children's Hospital Tirsova, Belgrade
  - Institute for Mother and Child Health Care of Serbia, Belgrade
  - University Clinical Centre Kragujevac, Kragujevac
  - University Clinical Centre Nis, Niš
  - Institute for Health Care of Children and Adolescents, Novi Sad
- Slovenia (2):
  - PeK - Dept. of Paediatric Endocrinology, Diabetes and Metabolism, Ljubljana
  - University Children's Hospital, Ljubljana
- South Africa (4):
  - Department of Peadiatrics CHBAH, Johannesburg, Gauteng
  - Dr JC van Dyk's Rooms, Pretoria, Gauteng
  - Dr Y Ganie's site, Mayville, KwaZulu-Natal
  - Dr K Pillay's site, Westville, KwaZulu-Natal
- South Korea (4):
  - Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do
  - Chungnam National University Sejong Hospital, Sejong-si
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
- Spain (4):
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela, A Coruña
  - H.Madrid Montepríncipe, Boadilla del Monte, Madrid
  - Hospital Madrid Montepríncipe, Boadilla del Monte, Madrid
  - Hospital Sant Joan de Déu, Esplugues de Llobregat
- Med. Kinder- und Poliklinik, Bern, Switzerland
- Thailand (9):
  - Ramathibodi Hospital - Ped-Endo and Metabolism, Ratchathewi, Bangkok
  - Ramathibodi Hospital - Ped-Endo and Metabolism, Bangkok, Ratchathewi
  - King Chulalongkorn Memorial hospital-Ped-Endocrinology, Bangkok
  - King Chulalongkorn Memorial hospital_Ped-Endocrinology, Bangkok
  - Phramongkutklao Hospital_Ped-Endo_Pediatrics, Bangkok
  - PMK - Paediatrics Endocrinology Centre, Bangkok
  - Siriraj Hospital_Dept of Paediatrics, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital_Pediatric Endocrinology, Chiang Mai
  - Srinagarind Hospital, Khon Kaen
- United Kingdom (8):
  - Addenbrooke's Hospital_Cambridge, Cambridge
  - Hull Royal Infirmary, Hull
  - Alder Hey Children's Hospital, Liverpool
  - Evelina Children's Hospital - St Thomas', London
  - Evelina London Children's Hospital, London
  - Royal Manchester Children's Hospital, Manchester
  - St George's Hospital, Tooting
  - St Georges Hospital, Tooting

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com